CLINICAL TRIAL: NCT05131672
Title: Operative Versus Nonoperative Treatment of Pediatric Medial Epicondyle Fractures (COMET Trial - Cast or Operation for Medial Epicondyle Fracture Treatment in Children)
Brief Title: Cast or Operation for Medial Epicondyle Fracture Treatment in Children
Acronym: COMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4916; 1U01AR079113 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-11-23 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Fracture Elbow
MeSH Terms: conditions — Elbow Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative reduction w/ fixation (Experimental): open reduction and internal fixation (ORIF)
  Interventions: Procedure: open reduction and internal fixation (ORIF)
- Non-operative immobilization (Active Comparator): immobilization in a cast without reduction
  Interventions: Procedure: cast immobilization

INTERVENTIONS:
Procedure: open reduction and internal fixation (ORIF) — open reduction and internal fixation with pin or screw fixation
  Arms: Operative reduction w/ fixation
Procedure: cast immobilization — immobilization in a cast without reduction
  Arms: Non-operative immobilization

SUMMARY:
This protocol describes a multicenter, prospective randomized superiority trial of medial epicondyle fracture treatments comparing functional outcomes between children treated with operative reduction and fixation or non-operative immobilization.

DETAILED DESCRIPTION:
INTRODUCTION

Fractures of the medial epicondyle are a common pediatric injury, with an estimated annual incidence of 40-60/100,000 per year. The typical mechanism is a fall onto an outstretched hand, creating a valgus load at the elbow leading to avulsion of the epicondyle from pull of either the flexor-pronator mass or ulnar collateral ligament. This injury is most frequent in children between the ages of 9 and 14, and is 4 times more likely in boys. Medial epicondyle fractures are associated with elbow dislocation in about 50% of cases, and ulnar nerve dysfunction is reported to occur nearly 10% of the time. No standard of care for medial epicondyle fractures exists, as similar outcomes have been demonstrated in observational studies with both operative and nonoperative treatment. Historically, most treatment has been nonsurgical, with immobilization of the injured elbow in a long-arm cast until healing. Increasingly, however, these injuries are being treated with surgical intervention, which in most cases consists of a single screw affixing the bony piece back to its donor site on the humerus.

No prospective studies have previously been performed evaluating the treatment of medial epicondyle fractures in children. All of the current literature on this issue has serious methodological limitations, such as lack of appropriate controls, retrospective assembly of cohorts, unstandardized assessment of outcomes, and irregular assessment of negative outcomes and adverse events. A 2009 systematic review of the literature identified 14 studies in which a comparison between operative and nonoperative treatment of medial epicondyle fractures in children or adolescents was performed. Of these, all were retrospective and observational in nature, with varying outcome measures utilized in the presentation of results.

There is considerable debate among clinicians as to the optimal management of medial epicondyle fractures, however, despite the lack of clear evidence of benefit, increasingly these injuries are being managed operatively. Explanations for the trend toward surgery focus on the athletic demands of children and adolescents, and the expectations of patients, parents, and coaches of early mobilization and return to sport. Because of the ongoing uncertainty as to best practice, a randomized trial is both ethical and indicated. High-quality data is necessary to better inform the decision regarding surgery and ensure both safe and effective treatment.

SAFETY OVERSIGHT

Safety oversight will be under the direction of a Data and Safety Monitoring Board (DSMB) composed of individuals with the appropriate expertise and knowledge of pediatric orthopaedic surgery usually obtained via an accredited pediatric orthopaedic fellowship. Members of the DSMB should be independent from the study conduct and free of conflict of interest, or measures should be in place to minimize perceived conflict of interest. The DSMB will meet at least semiannually to assess safety data on each arm of the study. The DMSB will operate under the rules of an approved charter that will be written and reviewed at the organizational meeting of the DSMB. At this time, each data element that the DSMB needs to assess will be clearly defined. The DSMB will provide its input to NIAMS.

QUALITY ASSURANCE AND QUALITY CONTROL

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted and data are generated and biological specimens are collected, documented (recorded), and reported in compliance with the protocol, International Conference on Harmonisation Good Clinical Practice (ICH GCP), and applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP)).

The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

DATA HANDLING AND RECORD KEEPING

DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site investigator. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

Clinical data and patient reported outcomes will be entered into REDCap, a 21 CFR Part 11-compliant data capture system provided by the DCRI. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.

STATISTICAL HYPOTHESES

• Primary Efficacy Endpoint(s):

The trial will employ a superiority framework. Specifically, the null hypothesis is that there is no difference in PROMIS UE (CAT) at 1 year between arms. The alternative hypothesis is that there is a difference between arms.

SAMPLE SIZE DETERMINATION

Sample size calculations were based on detecting a clinically meaningful difference in the Patient Reported Outcomes Measurement Information System (PROMIS) Upper extremity computer adaptive test (CAT) of 4 points. PROMIS measures use a T-score metric with a mean of 50 and standard deviation of 10 in a reference population. A sample size of 133 per am, assuming a two-sided type I error rate of 0.05, will provide 90% power to detect a difference between arms of 4 points.

To account for 20% lost-to-follow-up or missing data on the primary outcome at 12 months, we have inflated our sample size to 167 per arm, for a total target enrollment of 334.

A blinded sample size re-estimation based on the standard deviation of the primary outcome, after 50% of participants have completed the 6-month follow-up, will be performed.

POPULATIONS FOR ANALYSES

Primary analyses will be based on an Intention-to-treat (ITT) principle. A per-protocol analysis will be performed to assess the robustness of the ITT analysis. In the event of minimal (<5%) missing outcome data, primary analyses will be based on complete cases, reflecting a modified intent-to-treat analysis (mITT).

STATISTICAL ANALYSES

GENERAL APPROACH

Descriptive statistics will summarize all baseline variables by arm. Specifically, continuous variables will be summarized using mean and standard deviation, for normally distributed variables, and median and IQR, for non-normally distributed variables. Categorical variables will be summarized with frequency and percentages. There will be no formal hypothesis testing for comparison of baseline characteristics between treatment arms.

Primary analyses of the primary outcome at 1 year will be assessed with a two-sided type I error rate of 0.05. A false discovery rate (FDR) correction will be applied to analyses of all secondary outcomes to account for multiplicity.

ANALYSIS OF THE PRIMARY EFFICACY ENDPOINT(S)

Analysis for the primary aim will utilize a mixed effect model for the primary outcome, PROMIS Upper Extremity Function at 6 months, with a fixed effect for treatment arm and a random effect for site. Fixed effects will also include variables considered in the randomization (elbow dislocation status, age, sex) to control for imbalances in both the design and analysis. Incorporation of a random center effect will allow for separation of between site and within site variance components. Distributional assumptions will be assessed, and transformations or inclusions of higher order terms may be considered, as appropriate.

ANALYSIS OF THE SECONDARY ENDPOINT(S)

Secondary analyses will employ similar methods for all secondary continuous outcomes. Generalized linear mixed modeling approaches will be used for secondary binary and count outcomes, with appropriate link and distributional assumptions. All models will incorporate a random center effect and fixed effects for additional covariate considered in randomization, as described above.

Exploratory analyses may also consider trajectories of the primary outcome measured over time. Fixed effects for baseline PROMIS Upper Extremity Function, time, treatment arm, and the interaction will be included in a linear mixed effect model with random patient nested in center effects.

A False Discovery Rate (FDR) correction will be applied to all secondary analyses to account for multiplicity.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form by parent or legal guardian and signed assent form if participant is older than 12 years.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 7-17 years inclusive
4. Diagnosis of medial epicondyle fracture with any amount of displacement
5. Fracture is acute (occurred within 10 days of assignment of treatment arm)
6. Ability to take oral medication and be willing to adhere to the immobilization regimen

Exclusion Criteria:

1. Medial epicondyle fragment that is incarcerated within joint
2. Presence of other fractures about the ipsilateral elbow
3. Presence of pathologic fracture, open fracture
4. Have metabolic or neuromuscular diagnosis
5. Patient and parents are unable to adhere to procedures or complete follow-up due to insufficient comprehension of consent form or surveys or developmental delay.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 334 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
pediatric upper extremity function PROMIS computer adaptive test (PROMIS UE CAT) | 1 year follow-up
  functional and patient reported outcomes

SECONDARY OUTCOMES:
PROMIS UE Computerized Adaptive Test (CAT) | 6 weeks and 3, and 6 months
  functional and patient reported outcomes
Disabilities of the Arm, Shoulder and Hand (DASH) S/PA | 6 weeks and 3, and 6 months
  functional and patient reported outcomes
PROMIS Pain interference | 6 weeks, 3, 6, and 12 months
  functional and patient reported outcomes
Wong-Baker Faces Pain scores | 6 weeks, 3, 6, and 12 months
  functional and patient reported outcomes
Radiographic assessment of fracture healing | 3 months
  imaging
Number of revisions, refractures, re-reductions, and reoperations | within 1 year
  clinical outcomes
Estimated unit cost data for hospital and patient charges and costs | study duration
  cost data
PROMIS Global Health 7+2 | 3, 6, 12, 24, and 36 months
  functional and patient reported outcomes
Satisfaction questionnaire | 3,6, and 12 months
  functional and patient reported outcomes
Follow-up PROMIS Upper Extremity (UE) CAT | 12, 24 and 36 months
  functional and patient reported outcomes
Follow-up Disabilities of the Arm, Shoulder and Hand (DASH) S/PA | 12, 24 and 36 months
  functional and patient reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Janicki, MD, Principal Investigator — Ann and Robert H. Lurie Hospital Chicago
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States